CLINICAL TRIAL: NCT05167591
Title: Determination of Serum Paracetamol Concentration With an Electrochemical Measurement Tool From Blood and Saliva Samples in Patients Using Also Other Medication.
Brief Title: Detection of Paracetamol Concentration in Patients Using Regular Medication- a Validation Study for a Novel Technique
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: The design of the study is no longer relevant.
Sponsor: Johanna Kujala (Other)
Responsible Party: Sponsor-Investigator, Johanna Kujala, Sponsor-Investigator, Helsinki University Central Hospital
Organization: Helsinki University Central Hospital (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: FEPODPara2021-1
Record Dates: First submitted 2021-11-26; First posted 2021-12-22 (Actual); Last update posted 2024-03-06 (Actual); Status verified 2024-03

CONDITIONS: Pharmacokinetics
Keywords: Electrochemical; Paracetamol; Saliva; Fingerprick; Capillary sample; Acetaminophen

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Study group (Experimental): Measurements of paracetamol concentration
  Interventions: Diagnostic Test: Drug concentration measurement

INTERVENTIONS:
Diagnostic Test: Drug concentration measurement — Measurement of paracetamol concentration in capillary, venous plasma and saliva samples after standard premedication with paracetamol

SUMMARY:
Paracetamol intoxication is common, and concentration measurements are performed regularly. This research group is developing a fast bedside electrochemical analysis tool for paracetamol concentration measurement. This study will find out how this novel method performs in patients using other, confounding medication in detecting paracetamol concentration in capillary blood, venous plasma and saliva samples.

DETAILED DESCRIPTION:
Paracetamol concentration analysis is performed in 20 patients who will come to hospital for elective surgery. Inclusion criteria is a regular medication that continues over perioperative period.

Patients will be given standard premedication of paracetamol 1g perorally before surgery: this study does not affect standard surgical treatment.

Paracetamol concentration will be measured in venous plasma-, capillary blood-, and saliva samples before drug delivery and in recovery room after surgery using the novel electrochemical analysis tool and high-performance mass spectrometry analysis as a reference. If needed, confounding medication is identified with large toxicologic mass spectrometry screen (UPLC-QTOF).

ELIGIBILITY:
Inclusion Criteria:

* informed consent
* Age 18-75 years
* American society of anesthesiologist classification 2-4
* planned elective surgery with standard premedication with paracetamol 1g po.
* at least one regular medication ongoing perioperatively
* eligibility for elective surgery
* negative pregnancy test in fertile women

Exclusion Criteria:

* American society of anesthesiologists classification 1
* contraindication for use of paracetamol as standard premedication
* pregnancy or lactation
* less than 3 months from previous drug research
* less than 3 months from previous blood donation
* anticipated difficult puncture of veins
* Body Mass Index lower than 18.5 or higher than 35

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2024-03-01 (Estimated); Primary Completion 2024-03-04 (Estimated); Study Completion 2024-03-04 (Estimated)

PRIMARY OUTCOMES:
No outcome for patients | 24 hours
  Comparison of paracetamol concentration (µmol/L) measurements in saliva-, plasma-, and capillary samples and between mass-spectrometry and electrochemical techniques.

CONTACTS AND LOCATIONS:
Overall Officials: Eija Kalso, Principal Investigator — University of Helsinki

IPD SHARING:
Plan to Share IPD: No